CLINICAL TRIAL: NCT02547545
Title: Macro-microscopic Syndrome Differentiation and Combination，Based on the "Chinese Medicine Clinical Phenotype" to Construct Breast Cancer Chemotherapy Risk Prediction Mathematical Model
Brief Title: Breast Cancer Chemotherapy Risk Prediction Mathematical Model
Acronym: BCCRPMM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Shaanxi Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2012LSK-021
Record Dates: First submitted 2015-09-07; First posted 2015-09-11 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- All: The side effects after chemotherapy were observed for all patients. Potential risk factors would be explored for the side effects such as chemotherapy realted vomit.

SUMMARY:
This is a cohort study. This study is to develop a predictive model of the side effects after chemotherapy, exploreing the potential risk factors of the side effects such as myelosuppression and chemotherapy realted vomit after the chemotherapy, so that it could help to alleviate patients' fear and anxiety about the side effects and the toxicity of chemotherapy. The potential risk factors were measured at baseline.

DETAILED DESCRIPTION:
Firstly, the investigator will extact the "macro" information about physical conditon, which comes from syndrome-constitutional differentiation in the light of Traditonal Chinease Medicine (TCM) theory. Then combined with the "micro" information about pathological and biological markers, "TCM clinical phenotype" is extracted by Text Mining, and shows the full picture of the clinical features of breast cancer, which will include most of risk factors related to occurrence of adverse of chemotherapy fo breast cancer patients to establish two corresponding quatitative databases. Furthermore, predictive models will be built according to the predictors selected from an analysis on new methods of econometrics-Granger causality and cointegration analysis between "TCM clinical phenotype" and adverse effects of chemotherapy. The research results will be used to establish effective predictive models to lay the foundation for optimizing individualized treatment program of breast cancer by TCM and Western medicine.

ELIGIBILITY:
Inclusion Criteria:

* THe female patients diagnosed with breast cancer by first histopathology;
* No tumor intervention therapy was conducted within one prior to the survey;
* KPS score≥60;
* Patients without sever idiopathic disease;
* Patients who can independently respond to a questionnaire
* Those who signed informed consent

Exclusion Criteria:

* Patients with sever idiopathic disease of the gastrointestinal tract, heart and blood vessels, liver,kidney, hematopoietic system, endocrine system and so on;
* Patients with previous or nogoing application of drugs affecting bone marrow hemoatopoietic function;
* Patients who complicated with a serious infection or severe liquid sickness;
* Psychiatric patients;
* Those who can not independently respond to a questionnaire

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: breast cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 795 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-03 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Myelosuppression of chemotherapy | 6 month
  Outcome is a bianry outcome, Yes or No variable. The primary outcome is wether the bone marrow suppression occurred or not for patients during the chemotherapy.

SECONDARY OUTCOMES:
Chemotherapy related vomit (side effects of chemotherapy) | 6 month
  Outcome is a bianry outcome, Yes or No variable. The secondary outcome is wether the chemotherapy realted vomit occurred or not for patients during the chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Liu, MD,PHD, Principal Investigator — +86 18991232576
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi'an, China